CLINICAL TRIAL: NCT01856361
Title: Ramipril for the Treatment of Oligospermia: A Double-Blind Randomized Control Trial
Brief Title: Ramipril for the Treatment of Oligospermia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not accrue as much as anticipated and the PI (Dabaja) is no longer at Weill Cornell.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1301013462
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Oligospermia; Teratospermia; Asthenozoospermia; Male Infertility
Keywords: Male infertility; Low sperm count; Poor sperm motility; Poor Sperm shape and morphology
MeSH Terms: conditions — Oligospermia; Teratozoospermia; Asthenozoospermia; Infertility, Male | interventions — Ramipril; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramipril (Experimental): The initial dose of ramipril will be 2.5 mg that will be started at visit 2, week zero of the study. The dose will be increased to 5 mg during visit 3, 4 weeks into the study, for a total of 32 weeks.
  Interventions: Drug: Ramipril
- Placebo (Sham Comparator): The placebo group will get a similar pill that will be started at visit 2, week zero of the study. Subjects will be asked to double the dose by taking two pills during visit 3, four weeks into the study, for a total of 32 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramipril — Angiotensin Converting Enzyme Inhibitor
  Other Names: Altace
  Arms: Ramipril
Drug: Placebo — Placebo pill that will match the treatment pill
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial to evaluate the effect of ramipril in stimulating and promoting sperm production in men with low sperm count. Ramipril is an Angiotensin Converting Enzyme Inhibitor (ACEI) currently used to treat high blood pressure. However, previous studies have shown that this class of medications can improve sperm parameters. The purpose of this study is to evaluate the efficacy of ramipril compared to placebo (Substance That is not known to have treatment effect), in improving sperm density in infertile men with documented low sperm count. This study will help us identify subjects that might benefit from treatment with this medication, and the effect it will have on sperm count, shape, and motility.

DETAILED DESCRIPTION:
Approximately half of all infertility problems are caused by male factors. These men account for 17% of patients at the primary health care level that seek help for infertility. Oligospermia (Low sperm count) of unknown cause occurs in up to 60% of men with unexplained infertility. Certain group of patients with oligospermia can father children, but those with infertility have long posed a major therapeutic challenge. A variety of empirical non-specific treatments have been used, in attempt to improve their semen characteristics and fertility. In the past, androgens were suggested as a treatment; however, exogenous testosterone was found to exert negative feedback on the pituitary-gonadal axis and thereby suppresses Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) secretion then adversely affects sperm production. Other treatment modalities like clomiphene citrate, tamoxifen, recombinant FSH, zinc, selenium, and L-carnitine have been tried with minimal success. In the present study we are proposing the use of an angiotensin converting enzyme inhibitor (ACEI) for the treatment of oligospermia. A recently published pilot study showed that the use of lisinopril improved sperm quantity and quality in oligospermic men. ACEI are inexpensive, safe, widely available, and, if effective in improving sperm production and quality, could avert couples from undergoing invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male partner of a couple presenting for infertility.
2. Moderate abnormalities of semen parameters (Mean sperm density <20 million, but ≥ 3 million/ml), and/or motility < 50%, and/or < 4% abnormal morphology on at least two separate occasions.
3. Age 18-45 years.
4. Normal renal function defined as Glomerular filtration rate > 90

Exclusion Criteria:

1. Patients that are currently taking thiazide, cyclosporin, lithium, and allopurinol or the use of these medications in the last 2 weeks.
2. The frequent use of NSAIDS (3 or more times a week).
3. Vasectomy reversal.
4. Regular use of tobacco products.
5. Mean white blood cell count >1 million/ml in the ejaculate.
6. Inability or unwillingness to participate in evaluations required by the study.
7. Potassium > 5.0.
8. Systolic blood pressure < 90 mmHg.
9. Currently use of ACEI

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Schlegel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, Department of Urology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Department of Urology Cornell — https://www.cornellurology.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramipril | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Sperm Density in Infertile Men With Documented Oligospermia.
Time Frame: 32 weeks
Population: Data was not collected on the 2 participants as the principal investigator on this trial moved to a different practice and thus the study terminated before any results could be analyzed.
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Total Motile Sperm Count(TMSC), Total Sperm Count, Sperm Motility, and Morphology in the Ejaculate.
Description: The efficacy of ramipril in improving total sperm count will be evaluated, as well as, improving sperm motility, and morphology.
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pregnancy Rate
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hormonal Profile
Description: LH, FSH, serum testosterone, prolactin
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Seminal Angiotensin II and Serum Bradykinin Levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ramipril | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes